CLINICAL TRIAL: NCT06040827
Title: A Multicenter, Postmarket Surveillance Study of Subjects With the Canary canturioTM te Tibial Extension
Status: Recruiting | Type: Observational
Sponsor: Canary Medical (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Other Study IDs: PS220001
Record Dates: First submitted 2023-07-20; First posted 2023-09-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; Canary canturio™te; Zimmer Persona® Personalized Knee System; Zimmer Persona® Personalized Knee System with Canary canturioTM (CTE) tibial extension
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Group 1 (Test): Zimmer Persona® Personalized Knee System with Canary canturioTM (CTE) tibial extension
  Interventions: Device: Total Knee Arthroplasty
- Group 2 ( Control): Group 2 (Control): Zimmer Persona® Personalized Knee System with 14 mm +30 mm stem extension
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — The nature, severity, and frequency of safety risks (Adverse Events) in subjects with the Canary canturioTM te will be compared to those subjects with the legally marketed Zimmer Persona® Personalized Knee System with 14 mm x +30 mm stem extension within 5 years post-TKA.

SUMMARY:
The objectives of this prospective observational cohort study are to evaluate the safety, reliability, reproducibility, and accuracy of the Canary canturioTM te post-TKA.

DETAILED DESCRIPTION:
Group 1 (Test): Zimmer Persona® Personalized Knee System with Canary canturioTM (CTE) tibial extension Group 2 (Control): Zimmer Persona® Personalized Knee System with 14 mm +30 mm stem extension Safety Endpoint The nature, severity, and frequency of safety risks in subjects with the Canary canturioTM te will be compared to those subjects with the legally marketed Zimmer Persona® Personalized Knee System with 14 mm x +30 mm stem extension within 5 years post-TKA.

The safety endpoint is the percentage of patients that meet any of the following criteria within 5 years post-TKA:

* Revision (tibia only)
* Aseptic loosening
* Instability (or unrecognized septic loosening)
* Intra-operative fracture of bone or device
* Post-operative fracture of bone or device
* Radiologic changes including:
* Lytic lines (radiolucency greater than 2 mm in 2 or more zones)
* Focal lysis(progressive osteolytic lesion)
* Osteolysis (3mm in more than 1 zone)
* Device fracture or failure (tibia only)
* Cortical thickening or periosteal reactions

Secondary Endpoints

The secondary endpoints (for 5 years post-TKA) are:

Successful Data Collection

* Percent of days with step-count data transmitted
* Percent of days with one or more gait bouts triggered and transmitted
* Percent of days with qualified gait cycles >0 (applicable for walking speed, stride length, tibia ROM, functional knee ROM and cadence)
* Percent of days with step-count data transmitted and qualified gait cycles >0 (applicable for distance) Pain and Functional Performance
* Knee Injury and Osteoarthritis Outcome Score (KOOS - JR)
* Numeric Pain Rating Scale (NPRS)
* Quality-of-life- EQ-5D-5L

Effectiveness Endpoints (Reliability, Reproducibility, and Accuracy) The reliability, precision and accuracy of walking speed using measurements at 1 year and 2 years post TKA will be assessed with a cohort of 75 patients from Group 1 (with the CTE). Additionally, the reliability, precision and accuracy of all 7 gait parameters (walking speed, cadence, stride length, functional knee ROM, tibia ROM, step count and distance) using measurements at 1 year with 3 different walking speeds, will be assessed with a consecutive cohort of 25 patients from Group 1 in a gait lab.

ELIGIBILITY:
Inclusion

* Patient must be 18 years of age or older
* Patient qualifies for primary total knee arthroplasty based on physical exam and medical history, including diagnosis of severe knee pain and disability due to osteoarthritis, limited to:
* Mild or Moderate valgus, varus, or flexion deformities
* Patient must be willing and able to complete the protocol required follow-up
* Patient is indicated for a 58mm or 30mm tibial stem extension
* Patient has participated in the study-related informed consent process
* Patient is willing and able to provide written Informed Consent by signing and dating the IRB approved informed consent
* Patient has a platform-compatible personal computer located in their dwelling with appropriate wireless internet access and a USB port
* Independent of study participation, patient is a candidate for commercially available Persona Personalized Knee System implanted in accordance with product labeling

Exclusion

* Simultaneous bilateral TKA
* Staged bilateral TKA less than 6 months from indexed procedure
* Patient is a current alcohol or drug abuser
* Patient is known to be pregnant, breastfeeding, or considered a member of a protected class (e.g., prisoner, mentally incompetent, etc.)
* Patient has a psychiatric illness or cognitive deficit that will not allow proper informed consent and participation in follow-up program
* Patient has previous history of infection in the affected joint and/or a local or systemic infection that may affect the prosthetic joint
* Patient with mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions
* Patient with skeletal immaturity
* Patient has insufficient bone stock on femoral or tibial surfaces
* Patient with Neuropathic Arthropathy
* Patient has osteoporosis, or any loss of musculature or neuromuscular disease that compromises the affected limb
* Patient has severe instability secondary to the absence of collateral ligament integrity.
* Patient has a stable, painless arthrodesis in a satisfactory functional position
* Patient has rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
* Patient has a known or suspected sensitivity to one or more of the implant materials
* Patient is undergoing procedures or treatments using ionizing radiation
* Patients with known symptomatic foot, hip, or spinal injuries and/or conditions that could affect gait

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients indicated for a total knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 626 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | 5 years post TKA
  The nature, severity, and frequency of safety risks (Adverse Events) in subjects with the Canary canturioTM te will be compared to those subjects with the legally marketed Zimmer Persona® Personalized Knee System with 14 mm x +30 mm stem extension within 5 years post-TKA.

SECONDARY OUTCOMES:
Percent of days with step-count data transmitted | 5 years post TKA
  Successful Data Collection
Percent of days with one or more gait bouts triggered and transmitted | 5 years post TKA
  Successful Data Collection
Percent of days with qualified gait cycles >0 (applicable for walking speed meter/second, stride length meter, tibia ROM, functional knee ROM and cadence) | 5 years post TKA
  Successful Data Collection
Percent of days with step-count data transmitted and qualified gait cycles >0 (applicable for distance in meters) | 5 years post TKA
  Successful Data Collection
Knee Injury and Osteoarthritis Outcome Score (KOOS - JR) | 5 years post TKA
  Pain and Functional Performance
Numeric Pain Rating Scale (NPRS) | 5 years post TKA
  Pain and Functional Performance
Quality-of-life- EQ-5D-5L | 5 years post TKA
  Pain and Functional Performance

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Ozark Orthopaedics, Fayetteville, Arkansas
  - Foundation For Orthopaedic Research and Education, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - South Bend Orthopaedics, South Bend, Indiana
  - Cleveland Clinic, Cleveland, Ohio
  - JIS Research Institute, New Albany, Ohio
  - Carolina Orthopaedic & Neurosurgical Associates, Spartanburg, South Carolina